CLINICAL TRIAL: NCT07071909
Title: Immune Reconstitution Monitoring and Pneumococcal Vaccination (PCV-21) in Patients Treated With Chimeric Antigen Receptor T-Cells
Brief Title: Immune Reconstitution Monitoring and Pneumococcal Vaccination in Patients Treated With CAR-T Cells
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Funding unavailable
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: LCCC2337
Record Dates: First submitted 2025-07-08; First posted 2025-07-17 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Malignancy; Cancer; Hematological Malignancies; Lymphoma; Leukemia; Multiple Myeloma; Solid Tumor
Keywords: Chimeric antigen receptor (CAR)-T cell therapy; cell therapy; Chimeric antigen receptor (CAR)-T; infection; vaccine response
MeSH Terms: conditions — Neoplasms; Hematologic Neoplasms; Lymphoma; Leukemia; Multiple Myeloma; Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Commercial CAR-T (Experimental): Twenty subjects who are receiving commercial CAR-T for CD19 or BCMA.
  Interventions: Biological: Commercial CAR-T
- Investigational CAR-T (Experimental): Thirty subjects are 30 receiving investigational CAR-T through a University of North Carolina at Chapel Hill clinical trial.
  Interventions: Biological: Investigational CAR-T

INTERVENTIONS:
Biological: Commercial CAR-T — Twenty subjects will receive investigational CAR-T through a University of North Carolina at Chapel Hill clinical trial.
  Arms: Commercial CAR-T
Biological: Investigational CAR-T — Thirty subjects will receive investigational CAR-T through a University of North Carolina at Chapel Hill clinical trial.
  Arms: Investigational CAR-T

SUMMARY:
This is a prospective interventional study designed to investigate the effect of Immune Reconstitution clinic visits and pneumococcal vaccination (PCV-21) on infection risk, anti-infective prophylaxis adherence, and vaccine response in patients receiving CAR-T therapy following lymphodepletion. Fifty subjects (20 receiving commercial CAR-T for CD19 or BCMA and 30 receiving investigational CAR-T) will be enrolled. Subjects will attend Immune Reconstitution Clinic Visits at 3, 6, 9, and 12 months after CAR-T cell infusion. Subjects will be asked to provide blood samples at pre-defined intervals during CAR-T visits which will be assessed for immune composition, vaccine titers, viral titers, and immunoglobulins. Samples will be primarily used for study purposes. Leftover blood will be stored for up to five years after the last study visit and may be used for future research.

Vaccination against pneumococcal pneumonia will be offered at 6 months post-CAR-T infusion at the Immune Reconstitution Clinic Visit. Subjects will provide additional blood samples at 9- and 12 months post CAR-T infusion to assess anti-pneumococcal polysaccharide IgG antibodies to determine vaccine efficacy.

Long-term follow-up will continue for up to 24 months post-CAR-T infusion via medical chart abstraction.

This pilot study investigates immune reconstitution, infection risk, and vaccine response in patients receiving chimeric antigen receptor (CAR)-T cell therapy following lymphodepletion. Subjects will undergo lymphodepletion followed by CAR-T cell infusion will be included. The only additional treatment for subjects in this study is the PCV-21 pneumococcal vaccine. All CAR-T treatment procedures will adhere to the standard-of-care or the clinical trial protocol to which the subject is co-enrolled.

Subjects will provide blood samples at predefined intervals during CAR-T visits. These samples will be assessed for various laboratory studies, including blood counts, immune cell composition, viral titers, immunoglobulins, and microbiome composition.

Vaccination against pneumococcal pneumonia will be given 6 months post-CAR-T- T infusion. Subjects who opt for this vaccination will provide additional blood and blood samples at collected at 6, 9, and 12 months post-CAR-T infusion to assess anti-pneumococcal polysaccharide IgG antibodies. Long-term follow-up will continue for up to 24 months post-CAR-T infusion through medical chart abstraction

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent was obtained to participate in the study and HIPAA authorization for the release of personal health information.
2. The subject is willing and able to comply with study procedures based on the judgment of the investigator.
3. Age ≥ 18 years at the time of consent.
4. Planning to receive a commercial CD19 or BCMA-directed CAR-T therapy or investigational CD30 or solid tumor CAR-T therapy as a single infusion following lymphodepletion
5. Agree to provide blood samples as required by the protocol
6. Willing and able to provide access to immunization history
7. If receiving CAR-T as part of a clinical trial, must meet all eligibility criteria for that trial
8. Be willing to attend Immune Reconstitution Clinic Visits at 3, 6, 9, 12 months after CAR T-cell infusion
9. Be willing to receive PCV-21 vaccination at 6 months after CAR T-cell infusion.

Exclusion Criteria:

* None

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-01-20 (Actual); Primary Completion 2025-08-29 (Actual); Study Completion 2025-08-29 (Actual)

PRIMARY OUTCOMES:
Anti-pneumococcal antibody concentrations | Baseline, 3 and 6 months post vaccination
  Anti-pneumococcal titers will be measured in CAR-T patients to determine proportion of patients receiving either CD19 or BCMA-directed CAR-T vs CD30 or solid tumor CAR-T who respond to PCV21 vaccination.

SECONDARY OUTCOMES:
Number of reconstitution clinic visits | Up to 1 year
  Number of reconstitution clinic visits (PCP prophylaxis including sulfamethoxazole trimethoprim, pentamidine, daponse, or atovqaqune and HSV proprophylaxis including valacyclovir or acyclovir) compared to historic controls.
Difference in infection density | Up to 1 year
  Difference in infection density of patients within one year post CAR-T cell therapy infusion who attend Immune Reconstitution Clinic Visits compared to historic controls.

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Grover, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical trials at UNC Lineberger — http://unclineberger.org/patientcare/clinical-trials/clinical-trials